CLINICAL TRIAL: NCT06362746
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Trial of the Efficacy and Safety of a Single Bolus Administration of Non-immunogenic Recombinant Staphylokinase in Patients With Intermediate High-risk Pulmonary Embolism (FORPE-2)
Brief Title: Non-immunogenic Recombinant Staphylokinase vs Placebo in Patients With Intermediate High-risk Pulmonary Embolism
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Supergene, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FORPE-2
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Embolism
Keywords: Intermediate high-risk pulmonary embolism; Fibrinolysis; Recombinant Non-immunogenic Staphylokinase
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: At clinical sites patients will be equally randomized into two groups to receive non-immunogenic recombinant staphylokinase or placebo.
  Non-immunogenic recombinant staphylokinase or placebo will be administered intravenously at a dose of 15 mg as a single bolus for 10-15 seconds. All patients will be examined for 30 days.
Who Masked: Participant, Investigator
Masking Description: Neither patient nor investigator knows treatment assignment. All eligible patients will be randomized in two equal groups for administration of non-immunogenic recombinant staphylokinase or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-immunogenic recombinant staphylokinase (Experimental): lyophilisate for preparation of a solution for intravenous administration, 5 mg (745,000 IU) complete with a solvent. 15 mg (2,235,000 IU) - 3 vials, intravenously as a quick single bolus injection for 10-15 seconds, regardless of body weight.
  Interventions: Drug: Non-immunogenic recombinant staphylokinase
- Placebo (Placebo Comparator): 15 mg of placebo reconstituted in 15 ml of 0.9% solution of NaCl given as single i.v. bolus over 10-15 seconds
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Non-immunogenic recombinant staphylokinase — 15 mg of drug reconstituted in 15 ml of 0.9% solution of NaCl given as single i.v. bolus over 10-15 seconds
  Other Names: Fortelyzin®
  Arms: Non-immunogenic recombinant staphylokinase
Drug: Placebo — 15 mg of placebo reconstituted in 15 ml of 0.9% solution of NaCl given as single i.v. bolus over 10-15 seconds
  Arms: Placebo

SUMMARY:
Objective: to evaluate the efficacy and safety of the non-immunogenic recombinant staphylokinase with its single bolus administration in comparison with placebo in normotensive patients with intermediate high-risk pulmonary embolism (PE)

DETAILED DESCRIPTION:
For patients with massive PE thrombolysis can be life-saving and may reduce a pulmonary obstruction, pulmonary hypertension, and right ventricle dysfunction. Efficacy of the thrombolytic therapy has been proven in patients with high-risk pulmonary embolism accompanied by shock or systemic hypotension. However, the question of whether thrombolytic therapy can improve the clinical outcome of hemodynamically stable patients, i.e. with PE of intermediate high-risk, still remains controversial.

In PEITHO trial tenecteplase, administered as a single bolus at a dose of 30-50 mg depending on body weight was compared with a placebo in patients with intermediate high-risk PE with right ventricular dysfunction. Efficacy of tenecteplase was combined with a significant (6.3%) risk of hemorrhagic stroke, which did not allow tenecteplase to be included in the list of recommended thrombolytics for PE treatment.

PEITHO-3 trial has now begun, in which patients with intermediate high-risk PE are given a reduced dose of alteplase (0.6 mg/kg infusion with the total dose not exceeding 50 mg) compared with placebo.

Staphylokinase is a thrombolytic agent with high biological activity. Amino acid substitutions - including Lys74Ala, Glu75Ala, and Arg77Ala - resulted in a more than 200-times reduction in titres of neutralising antistaphylokinase IgGs in patients with ST-elevation myocardial infarction. In FORPE trial non-immunogenic recombinant staphylokinase was non-inferior as compared with alteplase in patients with high-risk massive PE.

The main objectives of this study: to assess the efficacy, safety and possible adverse events of the non-immunogenic recombinant staphylokinase with its single bolus administration in normotensive patients with intermediate high-risk PE in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over.
* Verified diagnosis of intermediate high-risk PE using CTPA, no more than two weeks from the symptoms onset.
* RV dysfunction, defined as a RV/LV ventricular end-diastolic diameter ratio more than 1.0 assessed by CTPA.
* Increased risk of early death or hemodynamic collapse, defined by one of the following criteria:

  1. systolic blood pressure less than 110 mm Hg, but not less than 90 mm Hg for more than 15 minutes;
  2. respiratory rate more than 20 per minute or SpO2 less than 90% without oxygen support;
  3. chronic heart failure with left ventricular ejection fraction less than 40%.
* Serum troponin I level more than 14 pg/mL in patients under 75 years, and more than 45 pg/mL in patients aged 75 years or older.
* Patient consent to use reliable contraceptive methods throughout the study and for 3 weeks after:

  * women who have a negative pregnancy test and use the following contraceptives: intrauterine devices, oral contraceptives, contraceptive patch, prolonged injectable contraceptives, double barrier method of contraception. Women who are not fertile can also take part in the study (documented conditions: hysterectomy, tubal ligation, infertility, menopause for more than 1 year);
  * men using barrier contraception. The study may also involve men who are not fertile (documented conditions: vasectomy, infertility).
* Availability of signed and dated informed consent of the patient to participate in the study.

Exclusion Criteria:

* High-risk PE with hemodynamic instability.
* Increased risk of bleeding:

  * extensive bleeding at present or within the previous 6 months;
  * intracranial (including subarachnoid) hemorrhage at present or in history;
  * hemorrhagic stroke within the last 6 months;
  * a history of diseases of the central nervous system (including neoplasms, aneurysms);
  * intracranial or spinal surgical interventions within the last 2 months;
  * major surgery or major trauma within the previous 4 weeks;
  * recent puncture of an incompressible blood vessel (eg, subclavian or jugular vein);
  * severe liver disease, including liver failure, cirrhosis, portal hypertension (including esophageal varices) and active hepatitis;
  * confirmed gastric or duodenal ulcer within the last 3 months;
  * neoplasm with an increased risk of bleeding;
  * simultaneous administration of Dabigatran without prior administration of idarucizumab;
  * arterial aneurysms, developmental defects of arteries / veins;
  * acute pancreatitis;
  * bacterial endocarditis, pericarditis;
  * suspicion of aortic dissecting aneurysm;
  * any other conditions, in the opinion of the investigator, associated with a high risk of bleeding.
* Lactation, pregnancy.
* Known hypersensitivity to the non-immunogenic recombinant staphylokinase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite of death from any cause or hemodynamic collapse or recurrent PE | within 30 days
  The efficacy is evaluated in terms of the number of death from any cause or hemodynamic collapse or recurrent PE

SECONDARY OUTCOMES:
Right/left ventricular (RV/LV) end-diastolic diameter ratio | within 24 hours
  The efficacy is evaluated in terms of the RV/LV end-diastolic diameter ratio according to echocardiography
RV/LV end-diastolic diameter ratio | within 24 hours
  The efficacy is evaluated in terms of the RV/LV end-diastolic diameter ratio according to computed tomography pulmonary angiography (CTPA)
RV/LV end-diastolic diameter ratio | within 30 days
  The efficacy is evaluated in terms of the RV/LV end-diastolic diameter ratio according to echocardiography
Right ventricular (RV) end-diastolic volume | within 24 hours
  The efficacy is evaluated in terms of the RV end-diastolic volume according to CTPA
Qanadli index | within 24 hours
  The efficacy is evaluated in terms of Qanadli index according to CTPA in points from 0 to 40, where 0 points - absence of thrombotic masses in the pulmonary artery, 40 points - complete occlusion of the pulmonary artery
Systolic pulmonary artery pressure | within 24 hours
  The efficacy is evaluated in terms of the systolic pulmonary artery pressure according to echocardiography
In hospital death from all causes (assessed up to day 7) | In hospital period (assessed up to day 7)
  The efficacy is evaluated in terms of the in hospital death from all causes (assessed up to day 7)
Death from all causes | within 30 days
  The efficacy is evaluated in terms of the death from all causes
Safety endpoint - hemorrhagic stroke | within 30 days
  The efficacy is evaluated in terms of the hemorrhagic stroke
Safety endpoint - BARC type 3 and 5 bleeding | within 30 days
  The efficacy is evaluated in terms of the Bleeding Academic Research Consortium definitions, where type 3a is an overt bleeding with hemoglobin drop of 3 to 5 g/dL and any transfusion with overt bleeding; type 3b is a bleeding requiring surgical intervention or intravenous vasoactive agents; type 3c is an intracranial hemorrhage; type 5 is fatal bleeding.
Safety endpoint - number and severity of adverse events (AEs) and serious AEs in organs and systems | within 30 days
  The efficacy is evaluated in terms of the number and severity of AEs and serious AEs in organs and systems

CONTACTS AND LOCATIONS:
Overall Officials: Sergey N. Tereschenko, MD, PhD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (24):
- Russia (24):
  - RZD Medicine hospital, Barnaul, Altayskiy Kray
  - V.F. Dolgopolov Vyselki Central District Hospital, Vyselki, Krasnodarskiy Kray
  - Asinovskaya District Hospital, Asino, Tomsk Oblast
  - Belgorod Regional Clinical Hospital of St. Joseph, Belgorod
  - Kuzbass Cardiology center, Kemerovo
  - Center of Neurology and Cardiology, Kirov
  - Regional Clinical Hospital №2, Krasnodar
  - Lipetsk City Hospital No. 4 "Lipetsk-Med", Lipetsk
  - F.I. Inozemtsev City Clinical Hospital, Moscow
  - Moscow Multidisciplinary Clinical Center "Kommunarka", Moscow
  - S.S. Yudin City Clinical Hospital, Moscow
  - V.M. Buyanov City Clinical Hospital, Moscow
  - S.P. Botkin City Clinical Hospital, Moscow
  - N.A. Semashko Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - N.N. Burdenko Penza Regional Clinical hospital, Penza
  - G.A. Zakharyin Clinical hospital №6, Penza
  - City Clinical Hospital №4, Perm
  - City Hospital No. 26, Saint Petersburg
  - City Hospital No. 15, Saint Petersburg
  - V.P. Polyakov Samara Regional Clinical Cardiology Dispensary, Samara
  - Tomsk regional cilinical hospital, Tomsk
  - Tver Regional Clinical Hospital, Tver'
  - Ufa Emergency City Hospital, Ufa
  - City Clinical Hospital of Emergency medicine №25, Volgograd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kirienko AI, Leontyev SG, Tereschenko SN, Yavelov IS, Shakhnovich RM, Erlikh AD, Talibov OB, Yarovaya EB, Semenov AM, Semenov MP, Ivanov SV, Beregovykh VV, Archakov AI, Markin SS; FORPE study group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with massive pulmonary embolism: a randomized open-label, multicenter, parallel-group, non-inferiority trial, FORPE. J Thromb Haemost. 2025 Feb;23(2):657-667. doi: 10.1016/j.jtha.2024.09.035. Epub 2024 Oct 23. PMID 39454884
- [Result] Leontyev SG, Yarovaya EB, Kutsenko VA, Ivlev OE, Soplenkova AG, Semenov AM, Semenov MP, Ivanov SV, Romashova YA, Markin SS. The Safety of Non-immunogenic Recombinant Staphylokinase in Elderly Patients With Massive Pulmonary Embolism: A Randomized Clinical Trial FORPE. Health Sci Rep. 2025 May 19;8(5):e70826. doi: 10.1002/hsr2.70826. eCollection 2025 May. PMID 40391253